CLINICAL TRIAL: NCT00786890
Title: A Survey to Evaluate the Cardiovascular Risk Status of Subjects With Pre-Diabetes in Hong Kong: The Joint Asia Diabetes Evaluation (JADE) Program Sub-study 2 (JADE-HK2)
Brief Title: A Survey to Evaluate the Cardiovascular Risk Status of Subjects With Pre-Diabetes in Hong Kong
Acronym: JADE-HK2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Other Study IDs: ADF-2008-2
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Prediabetes; Cardiovascular Risk Factors
Keywords: Prediabetes (IFG, IGT); Hong Kong Chinese; Cardiovascular risk factors
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- no treatment: observational, no treatment needed
  Interventions: Other: observational, no intervention needed

INTERVENTIONS:
Other: observational, no intervention needed — observational, no intervention needed

SUMMARY:
Hypothesis: A high cardiovascular risk is present in subjects with pre-diabetes in Hong Kong Chinese.

The investigators plan to assess Chinese subjects in Hong Kong who have pre-diabetes (impaired fasting glucose, IFG; or impaired glucose tolerance, IGT) based on oral glucose tolerance test (OGTT) on their cardiovascular risk status such as obesity, hypertension and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese with confirmed IFG or IGT by OGTT

Exclusion Criteria:

* Confirmed diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hong Kong Chinese with pre-diabetes
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk factors: anthroprometric parameters, blood pressure and lipid profiles | instant

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Institute of Diabetes and Obesity, Hong Kong, China